CLINICAL TRIAL: NCT04974645
Title: Pilot: Randomized Controlled Trial of an Digital Therapeutic Versus Education for the Management of Problematic Substance Use
Brief Title: Pilot: Digital Therapeutic vs Education for the Management of Problematic Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Collaborators: Stanford University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62053
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Use Disorder (AUD); Substance Use Disorders
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-SUDs (Experimental): Woebot (W-SUDs), a Conversational Agent (CA) instantaneously available 24 hours per day, 7 days per week, 'checks in' with users. Using conversational tones, it encourages mood tracking and delivers general psychoeducation as well as tailored empathy, cognitive behavior therapy (CBT)-based behavior change tools, and behavioral pattern insight. Woebot's app-based platform and user-centered design philosophy makes it an optimal modality for Substance Use Disorders (SUD) treatment delivery. It offers immediate, evidence-based tailored support in the patient's peak moment of craving.
  Interventions: Device: W-SUDs
- Digitally-delivered Psychoeducation (Other): Psychoeducation digitally delivers weekly fact sheets that include information on:
  1. Alcohol-specific topics;
  2. Drug-specific topics;
  3. General addiction topics;
  4. Statistics relating to alcohol and substance use.
  Interventions: Other: Digitally-delivered Psychoeducation

INTERVENTIONS:
Device: W-SUDs — Woebot (W-SUDs) is an automated conversational agent, available through a smartphone application, that delivers evidence-based psychotherapeutics, empathy, and emotional health psychoeducation.
  Arms: W-SUDs
Other: Digitally-delivered Psychoeducation — A form of psychoeducation for those seeking treatment for their alcohol and/or substance use concern. Psychoeducation is commonly provided for those with substance use. Psychoeducation in substance use is intended to increase the users' knowledge of their substances of use, and effects on the body, behaviors, and consequences. The recipient of psychoeducation is expected to increase their own awareness of their substance use and ideally incorporate this newfound knowledge when making changes to their substance use. The information provided in this group are from factsheets found on NIAAA, NIDA, and CDC web pages.
  Arms: Digitally-delivered Psychoeducation

SUMMARY:
Prior to launching a randomized controlled trial, this pilot study will investigate the feasibility and acceptability of the administration of a diagnostic interview and collection of a biomarker test, as well as engagement and preliminary efficacy with W-SUDs and the education arm, among a sample of adults who screen positive for problematic substance use.

ELIGIBILITY:
Inclusion Criteria:

1. Have a smartphone
2. Endorse a substance use concern
3. Be between 18 and 65 years of age
4. Be available and committed to engage with the Woebot app
5. Be literate in English.(This is required for inclusion because all materials will be in English).

Exclusion Criteria:

1. Pregnancy (as W-SUDs will not be specifically developed to address the unique needs of this population)
2. Suicide attempt within the past year (12 months)
3. Symptoms of severe drug/alcohol history: History of delirium tremens; Experiencing hypertension, drenching sweats, seizures or confusion after stopping alcohol or drugs; Liver trouble (cirrhosis or hepatitis); Convulsions or GI bleeding due to drug/alcohol use
4. Opioid overdose within the past year (12 months)
5. Opioid misuse without medication-assisted treatment
6. Not residing in the U.S.
7. Ever used Woebot

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Woebot Health, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Education: Education digitally delivers weekly fact sheets that include information on:
  1. Alcohol-specific topics;
  2. Drug-specific topics;
  3. General addiction topics;
  4. Statistics relating to alcohol and substance use.
  Education: The education arm will receive digitally delivered psychoeducation for those seeking treatment for their alcohol and/or substance use concern. Psychoeducation is commonly provided for those with substance use. Psychoeducation in substance use is intended to increase the users' knowledge of their substances of use, and effects on the body, behaviors, and consequences. The recipient of psychoeducation is expected to increase their own awareness of their substance use and ideally incorporate this newfound knowledge when making changes to their substance use. The information provided in this group are from factsheets found on NIAAA, NIDA, and CDC web pages.
Period: Overall Study
Arm/Group | W-SUDs | Education
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | W-SUDs | Education | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.5) | 43.3 (7.8) | 43.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 7 | 15
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Gender [Count of Participants; unit: Participants]
  Man | 7 | 3 | 10
  Woman | 2 | 7 | 9
  Genderqueer/Gender Non-conforming | 1 | 0 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 8 | 10 | 18
  Gay/Lesbian | 2 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Married/Partnered/Cohabitating | 7 | 2 | 9
  Divorced/Separated | 1 | 2 | 3
  Widowed | 0 | 1 | 1
  Single | 2 | 5 | 7
Highest Level of Education [Count of Participants; unit: Participants]
  Secondary/High School | 7 | 4 | 11
  College/University | 2 | 4 | 6
  Graduate/Postgraduate | 1 | 2 | 3
Therapy Experience [Count of Participants; unit: Participants]
  Experience in therapy | 6 | 8 | 14
  No therapy experience | 4 | 2 | 6
Past 30 Day Therapy [Count of Participants; unit: Participants]
  Outpatient Services | 2 | 2 | 4
  Multiple (self-help, outpatient, residential/inpatient/detox) | 0 | 1 | 1
  None | 6 | 5 | 11
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Substance Use Occasions
Description: Change in number of substance use occasions in the past 30 days
Time Frame: Change from Baseline to Mid-Treatment at 4 weeks; Change from Baseline to Post-treatment at 8 weeks; Change from Baseline to 1-Month Follow-up at 12 weeks
Measure: Mean (Standard Deviation); unit: occasions
Groups:
- Digitally-delivered Psychoeducation: Psychoeducation digitally delivers weekly fact sheets that include information on:
  1. Alcohol-specific topics;
  2. Drug-specific topics;
  3. General addiction topics;
  4. Statistics relating to alcohol and substance use.
  Psychoeducation: A form of psychoeducation for those seeking treatment for their alcohol and/or substance use concern. Psychoeducation is commonly provided for those with substance use. Psychoeducation in substance use is intended to increase the users' knowledge of their substances of use, and effects on the body, behaviors, and consequences. The recipient of psychoeducation is expected to increase their own awareness of their substance use and ideally incorporate this newfound knowledge when making changes to their substance use. The information provided in this group are from factsheets found on NIAAA, NIDA, and CDC web pages.
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
occasions
  Baseline to Mid-treatment at 4 weeks | -0.6 (18.3) | -7.2 (28.3)
  Baseline to Post-treatment at 8 weeks | -3.9 (20.6) | -6.7 (27.8)
  Baseline to 1-month Follow-up at 12 weeks | -4.9 (21.3) | -6.6 (37.8)

2. Secondary Outcome: Past Month Average Days Per Week of Drinking Alcohol
Description: Assessed with the Quick Drinking Screen (QDS), a measure of alcohol consumption. The QDS is a brief self-report measure used to assess average alcohol consumption over a specified time period (in the present study it was the past 30 days). The QDS collects drinking data for three variables including number of days drinking, number of standard drinks per drinking day, and number of binge/risky drinking days. Binge/risky drinking days is defined as days when they have had 5 or more standard drinks (for men) or 4 or more standard drinks (for women).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: days per week
Groups:
- Digitally-delivered Psychoeducation: Psychoeducation digitally delivers weekly fact sheets that include information on:
  1. Alcohol-specific topics;
  2. Drug-specific topics;
  3. General addiction topics;
  4. Statistics relating to alcohol and substance use.
  Digitally-delivered Psychoeducation: A form of psychoeducation for those seeking treatment for their alcohol and/or substance use concern. Psychoeducation is commonly provided for those with substance use. Psychoeducation in substance use is intended to increase the users' knowledge of their substances of use, and effects on the body, behaviors, and consequences. The recipient of psychoeducation is expected to increase their own awareness of their substance use and ideally incorporate this newfound knowledge when making changes to their substance use. The information provided in this group are from factsheets found on NIAAA, NIDA, and CDC web pages.
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
days per week
  Baseline to Mid-treatment at 4 weeks: Past month average days per week of drinking alcohol | -0.4 (0.9) | -2.4 (2.6)
  Baseline to Post-treatment at 8 weeks: Past month average days per week of drinking alcohol | -0.2 (0.8) | -1.6 (2.7)
  Baseline to 1-month Follow-up at 12 weeks: Past month average days per week of drinking alcohol | -0.6 (1.7) | -1.4 (2.7)

3. Secondary Outcome: Past Month Average Standard Drinks in a Day
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
drinks per drinking day
  Baseline to Mid-treatment at 4 weeks: Past month average standard drinks in a day | 1.6 (2.5) | -1.0 (3.0)
  Baseline to Post-treatment at 8 weeks: Past month average standard drinks in a day | -0.3 (0.8) | -1.1 (2.8)
  Baseline to 1-month Follow-up at 12 weeks: Past month average standard drinks in a day | -2.4 (6.0) | -0.8 (3.0)

4. Secondary Outcome: Past Month Number of Binge Days
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
days
  Baseline to Mid-treatment at 4 weeks: Past month number of binge days | 4 (11.6) | -1.3 (9.0)
  Baseline to Post-treatment at 8 weeks: Past month number of binge days | 2.0 (9.9) | -7.4 (9.6)
  Baseline to 1-month Follow-up at 12 weeks: Past month number of binge days | -3.7 (7.3) | -4.1 (11.1)

5. Secondary Outcome: Past Month Average Standard Drinks in a Week
Description: Assessed with the Quick Drinking Screen (QDS), a measure of alcohol consumption. The QDS is a brief self-report measure used to assess average alcohol consumption over a specified time period (in the present study it was the past 30 days). The QDS collects drinking data for three variables including number of days drinking, number of standard drinks per drinking day, and number of binge/risky drinking days. Binge/risky drinking days is defined as days when they have had 5 or more standard drinks (for men) or 4 or more standard drinks (for women). Number of standard drinks per week is calculated by multiplying number of standard drinks per day in the past month and number of binge days per month.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
drinks per week
  Baseline to Mid-treatment at 4 weeks: Past month average standard drinks in a week | 8.2 (19.2) | -8.0 (14.2)
  Baseline to Post-treatment at 8 weeks: Past month average standard drinks in a week | -2.3 (4.1) | -6.7 (13.8)
  Baseline to 1-month Follow-up at 12 weeks: Past month average standard drinks in a week | -10.3 (17.2) | -4.6 (16.2)

6. Secondary Outcome: Short Inventory of Problems- Alcohol and Drugs (SIP-AD)
Description: The SIP-AD assesses substance use problems in the past 30 days. The scored variables, total scores and 15-item mean, summarize consequences of alcohol and drug use. Scores range from 0-45, where greater scores indicate greater substance use problems.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline to Mid-Treatment at 4 weeks | -7.6 (9.2) | -1.1 (10.5)
  Baseline to Post-treatment at 8 weeks | -7.4 (8.4) | -4.0 (13.3)
  Baseline to 1-Month Follow-up at 12 weeks | -9.6 (8.1) | -4.4 (12.7)

7. Secondary Outcome: Craving Ratings
Description: Self-reported ratings of craving intensity. Craving is assessed with a single question, "In the past 7 days, how much were you bothered by cravings or urges to drink alcohol or use drugs?". The question is rated on a scale of 0 to 4 where 0 = not at all, 1 = a little bit, 2 = moderately, 3 = quite a bit, and 4 = extremely. Greater scores indicate a more intense urge to use.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline to Mid-Treatment at 4 weeks | -0.1 (0.7) | 0.0 (1.2)
  Baseline to Post-treatment at 8 weeks | -0.3 (0.7) | -0.1 (1.4)
  Baseline to 1-Month Follow-up at 12 weeks | -0.3 (0.8) | -0.3 (1.3)

8. Secondary Outcome: Working Alliance Inventory (WAI-SR)
Description: Measure of working alliance. A measure of therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Task, goal, and bond subscales scores range from 5-20, with higher scores indicating greater alliance. The present study utilized the validated 12-item Short-Revised version (WAI-SR) with minor changes to language, replacing "therapist" with "Woebot".
Time Frame: Difference between Mid-treatment at 4 weeks and Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs
Number analyzed (Participants) | 8
score on a scale
  Goal | 0.14 (4.56)
  Task | 0.57 (5.03)
  Bond | 1.57 (3.95)

9. Secondary Outcome: Stanford Presenteeism Scale (SPS-6)
Description: Measure of the effects of substance use on productivity. The SPS-6 is a 6-item self-report measure used to assess perceptions of the effects of substance use on past 2-week work productivity. Response options range from strongly disagree (1) to strongly agree (5). Total scores range from 6 to 30, where higher scores indicate higher presenteeism.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 6 | 6
score on a scale | 2.3 (3.7) | 2.7 (3.4)

10. Secondary Outcome: Thoughts About Abstinence (TAA)
Description: Modified for alcohol and substances. 5-item questionnaire assessing desire to quit, expected success at quitting, expected difficulty of quitting, and confidence in ability to quit. Each item is rated on a scale of 1 to 10 where 1 is the lowest (desire, expectation, confidence) and 10 is the highest (desire, expectation, confidence).
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 8 | 10
score on a scale
  Desire to quit | -0.8 (1.4) | 1.4 (2.0)
  Perceived success in quitting | 0.4 (2.3) | -0.8 (1.9)
  Difficulty in staying quit | 0.6 (3.7) | -0.6 (2.8)

11. Secondary Outcome: CAIR Pandemic Impact Questionnaire (C-PIQ)
Description: Assesses impact of the COVID-19 pandemic in terms of exposure to stressors, mental health impact and growth. Exposure domain total scores range from 0-15, with higher scores indicating greater exposure. Impact domain total scores range from 0-23, where greater scores are related to greater impact.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 8 | 10
score on a scale
  Exposure | -1.1 (1.7) | 0.1 (0.6)
  Impact | -2.8 (2.4) | -1.3 (1.3)

12. Secondary Outcome: Patient Health Questionnaire (PHQ-8)
Description: Measure of depression severity. An 8-item abbreviated version of the PHQ-9 used to assess mood symptoms. The PHQ-8 excludes an item assessing suicidality. Items are rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day"). Total score between 0-24, with higher scores indicating greater severity of depression symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline to Mid-treatment at 4 weeks | -3.9 (6.3) | -2.0 (5.2)
  Baseline to Post-treatment at 8 weeks | -1.9 (4.4) | -1.2 (6.5)
  Baseline to 1-month Follow-up at 12 weeks | -1.4 (4.2) | -2.9 (5.2)

13. Secondary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: Measure of anxiety severity. A 7-item self-report measure used to assess the frequency and severity of anxious thoughts and behaviors over the past 2 weeks. Items are rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day").Total scores range from 0-21, where higher scores indicate greater severity of anxiety symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline to Mid-treatment at 4 weeks | -3.4 (4.2) | 0.6 (3.7)
  Baseline to Post-treatment at 8 weeks | -0.6 (2.2) | -0.2 (4.3)
  Baseline to 1-month Follow-up at 12 weeks | -2.7 (2.7) | 0.6 (3.3)

14. Secondary Outcome: Brief Situational Confidence Questionnaire (BSCQ)
Description: Measure of self-confidence. The 8-item BSCQ is a state dependent measure that assesses self-confidence to resist the urge to drink heavily or use drugs in a variety of situations. Each of the 8 scale situations consists of a 100-mm line, anchored by 0% ("not at all confident") and 100% ("totally confident") where clients are asked to indicate confidence on a scale from 0% to 100%. Higher scores are associated with greater confidence.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline to Mid-treatment at 4 weeks | 10.9 (9.5) | 20.7 (21.1)
  Baseline to Post-treatment at 8 weeks | 10.9 (12.8) | 18.9 (21.2)
  Baseline to 1-month Follow-up at 12 weeks | 9.2 (10.3) | 20.7 (20.9)

15. Secondary Outcome: Usage Rating Profile - Intervention (URPI)-Acceptability
Description: Measure of acceptability. A 9-item subscale that inquires about intervention acceptability. For the purposes of this study, an adapted 6-item version of the subscale was utilized. Items are rated on a 6-point Likert scale (1 = "strongly disagree" to 6 = "strongly agree"). Total acceptability scores range from 6-36, with higher scores indicating greater intervention acceptability.
Time Frame: Post-treatment (8 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 8 | 10
score on a scale | 24.1 (6.2) | 27.4 (8.4)

16. Secondary Outcome: Usage Rating Profile Intervention - Intervention (URPI)-Feasibility
Description: Measure of feasibility. A 6-item subscale that inquires about factors that impact treatment usage (i.e., intervention quality). Items are rated on a 6-point Likert scale (1 = "slightly disagree" to 6 = "strongly agree"). Total feasibility scores range from 6-36, with higher scores indicating greater intervention feasibility.
Time Frame: Post-treatment (8 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 8 | 10
score on a scale | 27.4 (5.3) | 34.2 (2.7)

17. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: Measure of satisfaction. An 8-item measure used to assess client's satisfaction with treatment on a 4-point scale. Example questions include, "How would you rate the quality of service you received"? and "Did you get the kind of service you wanted?" Total sums range from 8-32, with high scores indicating greater satisfaction with the W-SUDs mobile application.
Time Frame: Post-treatment (8 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 8 | 10
score on a scale | 23.4 (5.5) | 26.1 (6.6)

18. Secondary Outcome: Number of Participants Indicating Substance Use
Description: The alcohol use disorder and substance use disorder (non-alcohol) modules of the Mini-International Neuropsychiatric Interview (MINI) was used to assess a alcohol and substance use diagnosis.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 8 | 6
participants
  Alcohol (mild) | 0 | 1
  Alcohol (moderate) | 1 | 2
  Alcohol (severe) | 4 | 3
  Stimulant (severe) | 3 | 0
  Cocaine (moderate) | 0 | 1
  Hallucinogen (mild) | 0 | 1
  Inhalant (mild) | 1 | 0
  Cannabis (moderate) | 1 | 0
  Cannabis (severe) | 3 | 2
  Sedatives (mild) | 1 | 0
  Sedatives (severe) | 1 | 0
  Multiple Diagnoses | 5 | 2

19. Secondary Outcome: Number of Participants Providing PEth Sample Phosphatidylethanol (PEth)
Description: Phosphatidylethanol (PEth) is an alcohol biomarker, where a positive result is an indication of alcohol exposure during the 2-4 weeks prior to specimen collection. Participants were asked to complete PEth tests at Baseline and Post-treatment at 8 weeks.
Time Frame: Baseline and Post-treatment at 8 weeks
Measure: Number; unit: participants
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10 | 10
participants
  PEth completed at Baseline | 5 | 5
  PEth completed at Post-treatment at 8 weeks | 3 | 4

20. Secondary Outcome: Engagement With Control Condition
Description: Assessment of number of emails opened duration of study
Time Frame: Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: emails
Arm/Group | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 10
emails | 6.7 (2.4)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed at post-treatment and follow-up at 8-weeks and 12-weeks from baseline, respectively.
Description: Serious adverse events occurring during treatment were assessed for hospitalization related to substance use, suicide attempt, alcohol or drug overdose, and severe withdrawal (e.g., delirium tremens). Positive endorsements were followed up with questions about the timing, diagnosis, and resolution. If additional details were needed to determine whether the event was study related, a team member reached out to the participant.
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04974645/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04974645/SAP_002.pdf
  • Informed Consent Form (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04974645/ICF_001.pdf